CLINICAL TRIAL: NCT05202808
Title: RxSight Light Adjustable Lens (LAL) And Light Delivery Device (LDD) New Enrollment Study
Brief Title: RxSight Light Adjustable Lens and Light Delivery Device New Enrollment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RxSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSP-029
Record Dates: First submitted 2021-12-29; First posted 2022-01-24 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Aphakia; Cataract
Keywords: Light Adjustable Lens; LAL; Intraocular lens
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 2:1 to undergo experimental or control treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Light adjustable lens (LAL) and Light Delivery Device (LDD) (Experimental)
  Interventions: Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD)
- Control IOL (Active Comparator)
  Interventions: Device: Control IOL

INTERVENTIONS:
Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD) — Experimental treatment group will receive Light adjustable lens with Light delivery Device treatments
  Arms: Light adjustable lens (LAL) and Light Delivery Device (LDD)
Device: Control IOL — Control treatment group will receive a Control IOL
  Arms: Control IOL

SUMMARY:
The primary objective of this study is to conduct a post-approval study which compares the LAL to a monofocal control IOL for safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Must sign a written Informed Consent form and be willing to undergo cataract surgery for the implantation of an IOL with random assignment to either the RxSight LAL or the monofocal control IOL.
* Between the ages of 40 and 80 inclusive on the day the cataract surgery is performed.
* Willing and able to comply with the requirements for study specific procedures and visits.
* Able to complete a written questionnaire in English.

Exclusion Criteria:

* Pre-existing macular disease in either eye.
* Patients with sufficiently dense cataracts that preclude examination of the macula in either eye.
* History of uveitis in either eye.
* Evidence of ectasia in either eye.
* Previous intraocular surgery in either eye. Eyes with previous pterygium excision are permitted as long as the pterygium did not extend more than 2mm onto the cornea from the limbus.
* Subjects taking systemic medication that may increase sensitivity to UV light.
* Subjects taking a systemic medication that is considered toxic to the retina such as tamoxifen.
* History of ocular herpes simplex virus in either eye.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Vold Vision, Fayetteville, Arkansas
  - Reeve Woods Eye Center, Chico, California
  - The Eye Institute of West Florida, Largo, Florida
  - Newsom Eye, Sebring, Florida
  - Vance Thompson Vision, Alexandria, Minnesota
  - Vance Thompson Vision, Omaha, Nebraska
  - Center for Sight, Las Vegas, Nevada
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina
  - Vance Thompson Vision Clinic, Sioux Falls, South Dakota
  - Key-Whitman Eye Center, Dallas, Texas
  - Slade & Baker Vision, Houston, Texas
  - Texas Eye Research Center, Hurst, Texas
  - Focal Point Vision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Started | 335; 335 Eyes | 165; 165 Eyes
Completed | 332; 332 Eyes | 164; 164 Eyes
Not Completed | 3; 3 Eyes | 1; 1 Eyes
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL | Total
Number analyzed (Participants) | 335 | 165 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (6.9) | 67.1 (6.3) | 67.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227 | 106 | 333
  Male | 108 | 59 | 167
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 6 | 2 | 8
  Black or African American | 23 | 8 | 31
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Caucasian | 305 | 156 | 461
Region of Enrollment [Number; unit: participants]
  United States | 335 | 165 | 500

OUTCOME MEASURES:

1. Primary Outcome: Absolute Manifest Refraction Spherical Equivalent (MRSE) Compared Between the Two Study Groups, LAL and Control
Time Frame: Postop Month 6
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Number analyzed (Participants) | 332 | 164
Diopters | 0.210 (0.213) | 0.345 (0.265)

2. Primary Outcome: Absolute Manifest Cylinder (MRCYL) Compared Between the Two Study Groups, LAL and Control
Time Frame: Postop Month 6
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Number analyzed (Participants) | 332 | 164
Diopters | 0.262 (0.275) | 0.820 (0.554)

3. Secondary Outcome: Rate of Endothelial Cell Density Loss
Description: The median difference was compared against a 5% non-inferiority margin for endothelial cell density loss using a right-tail Mann-Whitney-Wilcoxon test with a significance level of 0.05.
Time Frame: Postop Month 6
Measure: Median (95% Confidence Interval); unit: percentage Endothelial Cell Change
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Number analyzed (Participants) | 185 | 97
percentage Endothelial Cell Change | 5.1 [3.8 to 7.0] | 4.9 [3.0 to 6.5]
Statistical Analysis 1: Comparison: Light Adjustable Lens (LAL) and Light Delivery Device (LDD) vs Control IOL; With a one-sided significance level of 0.05, a power of 0.80, a randomization ratio of 2:1, and then the Mann-Whitney-Wilcoxon asymptotic relative efficiency (A.R.E.) efficiency adjustment, the sample size per two-sample t-test is 192 LAL eyes and 96 Control eyes (total of 288), with an assumed dropout rate of 10%; Test type: Non-Inferiority — The endothelial cell loss (ECL) at 6 months was compared between the LAL and Control groups. The statistical hypothesis is: * H0: Median(LAL) - Median(control) ≥ 5% vs * Ha: Median(LAL) - Median(control) < 5% The median ECL for the LAL group is at most 5% higher than the median ECL for the Control group. The first co-primary safety endpoint is met if the median ECL of the LAL group is non-inferior to the Control group using a right-tail Wilcoxon test using a significance level of 0.05; p < 0.0001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.2, 90% CI 2-sided [-1.00 to 1.66]

4. Secondary Outcome: Rate of Retinal Findings
Description: Rate of retinal findings in the Light adjustable lens (LAL) and Light Delivery Device (LDD) treatment group only.
Time Frame: Postop Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Number analyzed (Participants) | 331
Participants | 0

5. Post Hoc Outcome: Odds and Odds Ratio of Achieving Uncorrected Distance Visual Acuity (UCDVA) 20/20 or Better at Postop Month 6 Compared Between the RxSight LAL and Control Group
Description: Success defined as UCDVA 20/20 or better, failure defined as UCDVA worse than 20/20. Odds defined as number of successes divided by number of failures.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Number analyzed (Participants) | 332 | 164
Participants
  UCDVA 20/20 or better | 274 | 83
  UCDVA worse than 20/20 | 58 | 81
Statistical Analysis 1: Comparison: Light Adjustable Lens (LAL) and Light Delivery Device (LDD) vs Control IOL; Test type: Other; Odds Ratio (OR) = 4.61, 95% CI 2-sided [2.97 to 7.15] — Light adjustable lens (LAL) and Light Delivery Device (LDD) group is the numerator and Control group is the denominator. At Month 6, the odds of achieving UCDVA of 20/20 or better were 4.61 times greater for the LAL group than the Control group

6. Post Hoc Outcome: Odds and Odds Ratio of Achieving 0.5 Diopters or Less of Absolute MRCYL Compared Between the RxSight LAL and Control Group
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Number analyzed (Participants) | 332 | 164
Participants
  Absolute MRCYL 0.50 D or less | 307 | 61
  Absolute MCRYL worse than 0.50 D | 25 | 103
Statistical Analysis 1: Comparison: Light Adjustable Lens (LAL) and Light Delivery Device (LDD) vs Control IOL; Test type: Other; Odds Ratio (OR) = 20.74, 95% CI 2-sided [12.05 to 36.14] — Light adjustable lens (LAL) and Light Delivery Device (LDD) group is the numerator and the Control group is the denominator. The odds of achieving Absolute MRCYL of 0.5D or less was 20.74 for the LAL group versus the Control group at month 6

7. Post Hoc Outcome: Odds and Odds Ratio of Achieving Simultaneous Absolute Manifest Refraction Spherical Equivalent (MRSE) and Absolute Manifest Cylinder (MRCYL) of 0.50 D or Less at Postop Month 6 Compared Between the RxSight LAL and Control Group
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Number analyzed (Participants) | 332 | 164
Participants
  Simultaneous absolute MRSE and absolute MRCYL of 0.50 D or less | 291 | 54
  Simultaneous absolute MRSE and absolute MRCYL worse than 0.50 D | 41 | 110
Statistical Analysis 1: Comparison: Light Adjustable Lens (LAL) and Light Delivery Device (LDD) vs Control IOL; Test type: Other; Odds Ratio (OR) = 14.46, 95% CI 2-sided [8.89 to 23.57] — Light adjustable lens (LAL) and Light Delivery Device (LDD) group is the numerator and the Control group is the denominator. The odds of achieving simultaneous Absolute MRSE and MRCL of 0.5 D or less was 14.46 in the LAL group vs. Control at month 6

ADVERSE EVENTS:
Time Frame: 6 months
Description: Non-serious, ocular AEs are being reported for study eyes only.
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
All-Cause Mortality (participants affected / at risk) | 0/335 | 0/165
Serious Adverse Events (participants affected / at risk) | 7/335 | 2/165
Other Adverse Events (participants affected / at risk) | 71/335 | 26/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) (N=335) | Control IOL (N=165)
Secondary Surgical Intervention: Intraocular Lens Exchange (Surgical and medical procedures) | 0 (0) | 1 (1)
Secondary Surgical Intervention: Iris Repositioning following prolapse (Surgical and medical procedures) | 1 (1) | 0 (0)
Secondary Surgical Intervention: Study Eye, Selective Laser Trabeculoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Secondary Surgical Intervention: Non-Study Eye Intraocular Lens Exchange (Surgical and medical procedures) | 1 (1) | 0 (0)
Non-Study Eye, Full Thickness Macular Hole (Eye disorders) | 1 (1) | 0 (0)
Secondary Surgical Intervention: Non-Study Eye, Macular Hole Repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Inpatient hospitalization following Hip Replacement Surgery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inpatient hospitalization for Ventral Hernia Repair Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Inpatient hospitalization due to Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Inpatient hospitalization due to Salmonella Infection (Infections and infestations) | 1 (1) | 0 (0)
Inpatient hospitalization due to Obstruction of Gallbladder (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) (N=335) | Control IOL (N=165)
Allergic Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Amaurosis Fugax (Eye disorders) | 1 (1) | 0 (0)
Anterior Chamber Inflammation (Eye disorders) | 6 (7) | 6 (7)
Blepharoplasty (Surgical and medical procedures) | 1 (2) | 0 (0)
Blurry Vision (Eye disorders) | 1 (1) | 0 (0)
Clinically significant cystoid macular edema (Eye disorders) | 2 (2) | 4 (4)
Conjunctival Cyst (Eye disorders) | 0 (0) | 1 (1)
Corneal Abrasion (Eye disorders) | 4 (4) | 1 (1)
Cystoid Macular Edema (Eye disorders) | 0 (0) | 1 (1)
De-centered optic (Eye disorders) | 0 (0) | 1 (1)
Dot Hemorrhage (Eye disorders) | 1 (1) | 1 (1)
Epithelial Defect (Eye disorders) | 0 (0) | 1 (1)
Hypertensive Retinopathy (Eye disorders) | 1 (1) | 2 (2)
Iritis (Eye disorders) | 2 (2) | 1 (1)
Keratoconjunctivitis Sicca, not specified as Sjogrens (Eye disorders) | 2 (2) | 1 (2)
Corneal Erosion (Eye disorders) | 1 (1) | 0 (0)
Corneal Edema (Eye disorders) | 2 (2) | 0 (0)
Conjunctivochalasis (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis Medicamentosa (Eye disorders) | 1 (1) | 0 (0)
Conjunctival Hyperemia (Eye disorders) | 1 (1) | 0 (0)
Visual Symptoms due to Concussion (Eye disorders) | 1 (1) | 0 (0)
Dot Hemorrhages and Microaneurysms (Eye disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 0 (0)
Dry Eye Syndrome (Eye disorders) | 7 (7) | 0 (0)
Epiretinal Membrane (Eye disorders) | 1 (1) | 0 (0)
Epithelial Basement Membrane Dystrophy (Eye disorders) | 1 (1) | 0 (0)
Erythropsia score 2 (red) any time after Week 3 or Erythropsia score 1 (pink) or 2 (red) at Month 6 (Eye disorders) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 2 (2) | 0 (0)
Headache (Eye disorders) | 1 (1) | 0 (0)
Hordeolum (Eye disorders) | 1 (1) | 0 (0)
Light Treatment Sensitivity (Eye disorders) | 1 (1) | 0 (0)
Loss of BCDVA of >= 10 letters (when compared to Preop and/or Postop Week 3 BCDVA) (Eye disorders) | 2 (2) | 4 (4)
Meibomian Gland Dysfunction (Eye disorders) | 0 (0) | 1 (1)
Ocular Allergies (Eye disorders) | 2 (2) | 0 (0)
Ocular Hypertension (Eye disorders) | 1 (1) | 0 (0)
Posterior Capsular tear (Eye disorders) | 1 (1) | 0 (0)
Posterior Vitreous Detachment (Eye disorders) | 2 (3) | 0 (0)
Raised IOP (Eye disorders) | 14 (14) | 5 (5)
Raised IOP >=10 mmHg above preop & >=25 mmHg (if present > Week 1), unrelated to mech. pupil. block (Eye disorders) | 3 (3) | 0 (0)
Rebound Iritis (Eye disorders) | 1 (1) | 0 (0)
Retinal Hole (Eye disorders) | 0 (0) | 1 (1)
Retinal Microaneurysm (Eye disorders) | 1 (1) | 0 (0)
Subconjunctival Abrasion with Hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Superficial Punctate Keratitis (Eye disorders) | 16 (16) | 2 (2)
Uveitis (Eye disorders) | 1 (1) | 1 (1)
Wound leak (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT05202808/Prot_SAP_000.pdf